CLINICAL TRIAL: NCT06317636
Title: Randomized, Double-blind, Placebo-controlled, Single-center, Noninferiority Trial of Ketamine Given During Sedation to Patients With Chronic Pain and Depression
Brief Title: Propofol-Enhanced Assessment of Ketamine for Chronic Pain and Depression
Acronym: PEAK
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theresa Lii, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 73487
Record Dates: First submitted 2024-02-27; First posted 2024-03-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Depression
Keywords: Chronic Pain; Depression; Ketamine; Propofol; Sedation; Psychotropic Drugs; Hypnotics and Sedatives; Dissociative Anesthetics
MeSH Terms: conditions — Chronic Pain; Depression | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Active Comparator): A one-time intravenous infusion of ketamine (0.5 mg/kg)
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): A one-time intravenous infusion of normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/kg ketamine infused intravenously over 40 minutes
  Other Names: Ketalar
  Arms: Ketamine
Drug: Normal saline — 0.9% normal saline infused intravenously over 40 minutes
  Other Names: 0.9% NaCl
  Arms: Saline

SUMMARY:
The goal of this clinical trial is to compare ketamine to a placebo when given as a single infusion during IV sedation in adults with chronic pain and depression. We do not know whether ketamine will be more effective than placebo under these circumstances.

This study aims to:

* Evaluate whether placebo is non-inferior to ketamine in treating chronic pain and depression, when delivered under propofol sedation
* Confirm that propofol sedation is a safe way to keep participants blinded to treatment
* Assess patients' comfort with the sedation process to improve future studies
* Explore whether patient expectations affects their pain and depression

Participants will:

* Need to qualify for the study based on stringent medical criteria
* Undergo sedation with propofol
* Randomly receive either a ketamine or a placebo (saline) infusion during sedation
* Complete several study assessments over 5-7 weeks

DETAILED DESCRIPTION:
Ketamine is a dissociative anesthetic that has been in clinical use for more than 50 years. In addition to its well-known anesthetic and pain-relieving properties, ketamine has been found to have fast-acting antidepressant effects in patients with depression. However, the mechanisms underlying ketamine's ability to treat chronic pain and depression are poorly understood. A most basic question regarding ketamine's therapeutic mechanism is still unresolved: do patients need to consciously experience and recall ketamine's acute dissociative effects to receive lasting analgesic and antidepressant benefits? In this clinical trial, participants will receive either ketamine or a placebo when they are under sedation with propofol. A n=6 pilot feasibility phase will precede the fully-powered n=34 randomized controlled trial.

Enrollment for the n=6 pilot phase is complete as of 6/19/2025.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old
* Comfortable speaking and writing in English
* Chronic pain present daily for at least 3 months
* Currently experiencing depression
* Able to comply with the study protocol and communicate with study personnel about adverse events and other clinically important information

Exclusion Criteria:

* Pregnant or breastfeeding
* One or more health conditions that makes study unsafe or unfeasible, determined by study physicians
* Regular use of medications that may have problematic interactions with the study drugs
* Participating in another clinical trial which may conflict with this one

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity in the past 24 hours | screening; 1, 7, 14, 21 and 28 days after treatment
  A numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain) over the past 24 hours will be used to assess pain intensity.

SECONDARY OUTCOMES:
Depression Severity and Blinding | screening; day of infusion pre-treatment; 7, 14, 21 and 28 days after treatment
  The 16-item Quick Inventory of Depressive Symptomatology Self-Report will be used to assess the severity of depressive symptoms. Items are self-rated on a 4-point scale tailored to each depression-related symptom. Higher total scores indicate greater depression symptom severity.
  Blinding will be assessed by asking participants to guess which treatment they received and rate their certainty on a simple 0-100 scale.

OTHER OUTCOMES:
Number and severity of adverse events related to sedation | during treatment; day of infusion post-treatment; 1, 7, 14, 21 and 28 days after treatment
  Adverse events (AEs) will be assessed through a combination of patient self-report, interviews by study staff, and surveillance of medical records by the research team. AEs will be graded by severity (1=mild, 2=moderate, 3=severe, 4=life threatening, and 5=death) and relatedness to the intervention (0=definitely unrelated, 1=unlikely, 2=possibly related, 3=probably related, 4 definitely related).
Side effects related to ketamine | day of infusion post-treatment; 1, 7, 14, 21 and 28 days after treatment
  The Ketamine Side Effect Tool (KSET) is a standardized questionnaire designed to systematically assess the side effects experienced during or after ketamine administration. It covers a range of potential adverse effects, including dissociative, cardiovascular, and psychotomimetic symptoms. Participants are asked to rate the severity of each adverse effect as 'Never', 'Mild', 'Moderate', or 'Severe'.
Proportion of participants who accurately recall intra-sedation events | day of infusion post-treatment
  Participants will be interviewed by study staff using the modified Brice Questionnaire, a set of questions asked in sequence to determine if the participant remembers anything between the time of induction and their awakening.
Participant expectations | screening; day of infusion post-treatment; 1, 7, 14, 21 and 28 days after treatment
  Expectations will be measured by asking participants to rate how effective they expect their treatment will be using a visual analog sliding scale from 0 ("Not effective at all") to 100 ("Completely effective"). They will then be asked to rate their level of confidence on a scale from 0 to 100%.
Pressure pain threshold | day of infusion pre-treatment; day of infusion post-treatment
  A pressure algometer device applied to the upper trapezius muscle will measure the pressure pain threshold by applying a controlled, gradually increasing force until the participant reports pain.
Mechanical temporal summation | day of infusion pre-treatment; day of infusion post-treatment
  Mechanical temporal summation will be measured by applying the blunt tip of a thin flexible filament to the back of the hand and the lumbar region. Participants will be asked report pain intensity on a sale from 0 to 100 after a single application and after 10 repeated applications.
Conditioned pain modulation | day of infusion pre-treatment; day of infusion post-treatment
  Conditioned pain modulation (CPM) measures the ability of the nervous system to inhibit a painful stimulus in the presence of another aversive stimulus. In this study, participants will immerse one hand in cold water and undergo pressure pain threshold measurements in the opposite trapezius muscle before, during, and after immersion.
Number of painful body regions | screening; day of infusion pre-treatment; day of infusion post-treatment; 1, 7, 14, 21 and 28 days after treatment
  The CHOIR Body Map is a visual tool that allows individuals to indicate the location(s) of their pain on a human body outline.
Pain interference | screening; day of infusion pre-treatment; 7, 14, 21 and 28 days after treatment
  The 8-item PROMIS Pain Interference Short Form assesses the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("Very Much"). Raw score totals are converted to standardized T-scores, with a higher T-score representing greater pain interference.
Change in pain medication utilization | 1, 7, 14, 21 and 28 days after treatment
  Participants are asked to rate how their pain medication usage has changed compared to before treatment
Physical function | screening; day of infusion pre-treatment; 7, 14, 21 and 28 days after treatment
  The 20-item PROMIS Physical Function Short Form assesses the ability to carry out physical tasks and activities in one's daily life. Items are self-rated on a 5-point scale ranging from 1 ("Unable to do") to 5 ("Without any difficulty"). Raw score totals are converted to standardized T-scores, with a higher T-score representing better physical function.
Sleep disturbance | screening; day of infusion pre-treatment; 7, 14, 21 and 28 days after treatment
  The 8-item PROMIS Sleep Disturbance Short Form assesses an individual's perception of their sleep quality. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("Very much"). Raw scores are converted to standardized T-scores, with higher a T-score representing more severe sleep disturbance.
Anxiety symptom severity | screening; day of infusion pre-treatment; 14 and 28 days after treatment]
  The 7-item Generalized Anxiety Disorder (GAD-7) Scale assesses the severity of anxiety symptomsover the past two weeks. Items are self-rated on a 4-point scale ranging from 0 ("Not at all") to 3 ("Nearly every day"), reflecting the frequency of symptoms. Higher total scores indicate greater anxiety symptom severity.
Peace of mind | screening; day of infusion pre-treatment; 7 and 28 days after treatment
  The 7-item Peace of Mind Scale assesses an individual's overall sense of inner calm and contentment. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("All of the time"). Higher total scores reflect a greater sense of peace of mind.
Emotion regulation | screening; day of infusion pre-treatment; 7 and 28 days after treatment
  The 10-item Emotion Regulation Questionnaire assesses individual differences in the habitual use of cognitive reappraisal and expressive suppression strategies. Items are self-rated on a 7-point scale ranging from 1 ("Strongly disagree") to 7 ("Strongly agree"). Higher scores on the cognitive reappraisal subscale indicate a greater tendency to reinterpret situations to manage emotions, while higher scores on the expressive suppression subscale indicate a greater tendency to inhibit outward emotional expression.
Anhedonia | screening; day of infusion pre-treatment; 14 and 28 days after treatment
  The 14-item Snaith-Hamilton Pleasure Scale measures an individual's capacity to experience pleasure from various activities over the past 2 weeks, the absence of which indicates anhedonia. Items are self-rated on a 4-point scale ranging from 0 ("Strongly disagree") to 3 ("Strongly agree"). Lower total scores indicate greater degree of anhedonia.
Enrollment rate | from date of opening enrollment to the date of consent from the last participant, assessed up to 60 months
  The total number of consented, eligible participants enrolled by the end of the study divided by the amount of time between date of opening enrollment and the date of consent from the last participant.
Consent fraction | from date of opening enrollment to the date of consent from the last participant, assessed up to 60 months
  The proportion of patients who are contacted by study staff for recruitment who provide written informed consent to study procedures.
Participant Experience Survey | through study completion, an average of 4 weeks
  Participants are asked at the end of the study to rate their experience with study procedures and to provide feedback for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Lii, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, study outcomes, and data dictionaries
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available upon request after publication of the trial's primary findings for up to 5 years.
Access Criteria: Researchers must submit a brief proposal and statistical analysis plan for review and approval by the investigators and execute a data sharing agreement.